CLINICAL TRIAL: NCT03945435
Title: Mechanisms of Exercise Resistance in Metabolic Disease
Status: Completed | Type: Observational
Sponsor: Joslin Diabetes Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-09
Record Dates: First submitted 2018-05-23; First posted 2019-05-10 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Impaired Glucose Tolerance
Keywords: Exercise; Cardiorespiratory Fitness; Skeletal Muscle; Angiogenesis
MeSH Terms: conditions — Glucose Intolerance; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum Skeletal Muscle
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal Glucose Tolerance: Blood glucose level of less than 140 mg/dL at the 2 hour timepoint.
- Impaired Glucose Tolerance: Blood glucose level of greater or equal to 140 mg/dL at the 2 hour timepoint.

SUMMARY:
This project will determine exercise capacity and molecular markers of the response to acute exercise in human subjects with impaired or normal glucose tolerance.

DETAILED DESCRIPTION:
Low exercise capacity is an early clinical marker of metabolic impairment that predicts type 2 diabetes (T2D) risk, as well as future co-morbidities and complications. Aerobic exercise training is the only effective treatment to increase exercise capacity and reduce metabolic risk. However, despite maintaining similar levels of physical activity, exercise capacity remains lower in people with impaired glucose tolerance and T2D, compared to those with normal glucose tolerance, suggesting "exercise resistance". The mechanisms of exercise resistance in metabolic disease are unknown. In preclinical studies, exercise-induced increases in circulating angiogenic markers and skeletal muscle capillary density predict improved exercise capacity with training. Furthermore, it was demonstrated that impaired glucose tolerance precedes exercise resistance and impaired exercise-induce angiogenesis in muscle. Based on these data, it was hypothesized that exercise resistance in human T2D is caused by an impaired angiogenic response to exercise, secondary to impaired glycemic control. This study will determine whether the angiogenic response to a single bout of exercise in human subjects is blunted in patients with impaired glucose tolerance (IGT), compared to those with normal glucose tolerance (NGT). Angiogenic potential will be measured using a novel in vitro assay developed to assess endothelial tube-formation induced by circulating serum angiogenic regulators following exercise. In addition, a novel exercise-activated signaling pathway in skeletal muscle that is predictive of exercise resistance in animal models was identified. A second aim of the proposed investigation is to determine the effect of impaired glucose tolerance on molecular signaling in response to exercise in skeletal muscle. This investigation represents a critical step in determining the mechanisms that contribute to low exercise capacity in individuals at risk for diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45, BMI 26-32 kg/m2, Sedentary Lifestyle

Exclusion Criteria:

* Type 1 or Type 2 diabetes, heart or lung disease, hypertension, contraindications to exercise testing, pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study population will be men and women from the Boston area
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
VO2peak | One week
  Cardiorespiratory Fitness

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Lessard, Ph.D., Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided